CLINICAL TRIAL: NCT01045278
Title: Hepatitis C in a Cohort of Patients With Maintenance Therapy for Opiate Dependence - Prevalence, Severity and Outcome of Antiviral Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EU-nr 2007-001130-13
Record Dates: First submitted 2009-09-11; First posted 2010-01-11 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-10

CONDITIONS: Hepatitis C
Keywords: Hepatitis C patients; Hepacivirus
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Pegylated interferon-alfa-2b and ribavirin — Pegylated interferon-alfa-2b 1.5 microg/kg subcutaneously once weekly plus weight based ribavirin 800-1200 mg PO for a variable period depending on their HCV genotype and response to treatment.

SUMMARY:
Hepatitis C is the leading cause of chronic liver disease in industrialized countries, and is the most common indication for liver transplantation. In the Western world, the absolute majority of cases of Hepatitis C Virus (HCV) infection are related to the use of injectable narcotic drugs. Most injecting drug users contract HCV infection within the first years after starting injecting drug use. The aim of this study is to study hepatitis C in a cohort of patients registered in clinics providing maintenance therapy for opiate dependence in three metropolitan areas of Sweden. The cohort is defined as all patients registered in these three clinics at the date of study initiation. The study contains four parts:

Part I: the first part of the study aims to evaluate the prevalence of HCV exposure in the cohort and the proportion of anti-HCV positive participants with chronic infection.

Part II: Patients with chronic HCV infection will be offered further investigation of chronic liver disease, including liver biopsy, for selection of candidates for antiviral therapy and identification of risk factors for development of severe liver disease.

Part III: Based on the results of these investigations, patients will be considered for antiviral therapy. Indications for such therapy will mainly be clinical and/or histological signs of chronic liver disease with fibrosis. All patients will receive weight-based doses of pegylated interferon-alfa-2b and ribavirin.

Part IV: Study of pharmacokinetic interactions between ribavirin and opiate substitution molecule (methadone or buprenorphine) in patients receiving antiviral therapy according to part III.

ELIGIBILITY:
Inclusion Criteria:

* Patients that meet all of the following inclusion criteria are eligible for part I of the study:

  1. Registered in a clinic providing maintenance therapy for opiate dependence at the date of study initiation.
  2. Written informed consent for part I of the study.
* Patients that meet all of the following inclusion criteria are eligible for part II of the study:

  1. Fulfilled part I
  2. Registered in a clinic providing maintenance therapy for opiate dependence at the date of study initiation.
  3. HCV-PCR positive.
  4. Written informed consent for part II of the study.
* Patients that meet all of the following inclusion criteria are eligible for part III of the study:

  1. Fulfilled part II
  2. Registered in a clinic providing maintenance therapy for opiate dependence at the date of study initiation.
  3. HCV-PCR positive.
  4. Written informed consent for part III of the study and able to adhere to dosing and visiting schedules.
  5. At least 6 months of uninterrupted maintenance therapy for opiate dependence.
  6. Treatment indication with at least one of the following:

     * Fibrosis/cirrhosis
     * Other HCV related disease/symptoms
     * Psychological indication
  7. For patients with cirrhosis, an ultrasound investigation should be performed within six months before study initiation, part III, (not showing signs of HCC).
  8. Use of adequate contraception during the treatment period and for six months after the completion of therapy (for all participants regardless of gender).

Exclusion Criteria:

* The presence of any of the following criteria will exclude the patient from participating in part III of the study:

  1. Pregnant women, women who plan to become pregnant, male patients whose partner wants to become pregnant, and breastfeeding women.
  2. Previous treatment for chronic hepatitis C with an antiviral or immunomodulating agent or with an interferon or ribavirin product, whether alone or in combination.
  3. Participation in another clinical drug trial.
  4. Coinfection with HBV or HIV
  5. Hemoglobin <120 g/L for females and <130 g/L for males.
  6. LPK <3,0 x 109/L
  7. Platelets <80 x 109/L
  8. Creatinin clearance <50mL/min
  9. Any of the following diseases considered to be a dominant cause of the patients chronic liver disease:

     * Hemochromatosis
     * Alpha-1 antitrypsin deficiency
     * Wilson's disease
     * Autoimmune hepatitis
     * Alcoholic liver disease
     * Non-alcoholic steatohepatitis (NASH)
     * Drug-related liver disease
  10. Active malignant disease or suspicion or history of malignant disease within five previous years (except for adequately treated basal cell carcinoma).
  11. Patients with organ transplants, except for corneal or hair transplant.
  12. Poorly controlled diabetes mellitus.
  13. Evidence of severe retinopathy or clinically relevant ophthalmological disorder in patients with diabetes mellitus or hypertension.
  14. Poorly controlled epilepsy.
  15. Thyroid dysfunction not adequately controlled
  16. Decompensated cirrhosis (Child-Pugh B-C).
  17. Treatment with immunomodulatory drugs (chronic systemic corticosteroids (equivalent to >10 mg prednisone/day), immunosuppressive drugs, chemotherapy) and/or treatment with herbal drugs for chronic hepatitis.
  18. Any other condition which in the opinion of the investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in and completing the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2008-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
To determine the completion rates of HCV treatment with pegylated interferon-alfa-2b and ribavirin in patients who are under opiate maintenance treatment and eligible for HCV therapy. | 14-72 weeks

SECONDARY OUTCOMES:
Prevalence of chronic HCV infection in the patient population eligible for part I in the study. | Screening visit (first visit of the study).
Clinical and histological characteristics of chronic hepatitis C. | Liver investigation visit (second visit of the study). No time frame specified in the protocol.
Prevalence of hepatic decompensation and cirrhosis/advanced liver disease. | Liver investigation visit (second visit of the study). No time frame specified in the protocol.
Risk factors for advanced liver disease. | Liver investigation visit (second visit of the study). No time frame specified in the protocol.
Proportion of sustained virological responders, defined as a plasma HVC RNA level below Lower Level of Quantification at 24 week post-treatment. | 24 weeks post-treatment.
Rates of relapse in opiate drug abuse. | Treatment period (14-72 weeks) and up till 24 weeks post-treatment.
Prevalence of depressive symptoms and assessment of quality of life before, under and after HCV treatment. | Treatment period (14-72 weeks) and up to 24 weeks post-treatment.
Potential pharmacokinetic interactions between ribavirin and methadone or buprenorphine. | Measured after 4 weeks treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Jerkeman, MD, Study Director — Skane University Hospital
Locations (1):
- Skåne university hospital, Malmo, Sweden